CLINICAL TRIAL: NCT05200351
Title: Equine-assisted Therapy for Therapy-resistant Adolescents With Autism Spectrum Disorders, a Replicated AB-design
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karakter Kinder- en Jeugdpsychiatrie (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 185-20 Pegasus; 636310020 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2021-12-17; First posted 2022-01-20 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Emotion Regulation; Autism Spectrum Disorder; Adolescent - Emotional Problem
MeSH Terms: conditions — Emotional Regulation; Autism Spectrum Disorder | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the five pre-defined baseline lengths (2-6 weeks) to increase the internal validity of the design with a 1:1 allocation using permuted blocks of random sizes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EAT Intervention (Experimental): 15 sessions of EAT
  Interventions: Behavioral: Equine assisted Therapy (EAT)

INTERVENTIONS:
Behavioral: Equine assisted Therapy (EAT) — 15 sessions of EAT will be given. Activities will be with or in the presence of the horse. There will be no horseriding.

SUMMARY:
The purpose of this study is to assess the (cost)effectivity of Equine assisted Therapy in adolescents with Autism Spectrum disorders.

DETAILED DESCRIPTION:
The study has a mixed-methods strategy consisting of three elements: a randomized, multiple-baseline single-case design (n=35), a qualitative study (n=8-10) and a cost-effectiveness study (n=6). After obtaining written informed consent, participants will be randomly assigned to one of the five pre-defined baseline lengths (2-6 weeks) to increase the internal validity of the design.

ELIGIBILITY:
Inclusion Criteria:

* between 11-18 years old;
* a clinical diagnosis of autism spectrum disorders according the Diagnostic and Statistical Manual of Mental Disorders 5 (DSM 5) as diagnosed by a Beroepen in de Individuele Gezondheidszorg (BIG) registered healthcare professional;
* insufficient emotion regulation after regular therapy for at least 1,5 years as indicated by a score above clinical cut-off (T-score = 65) on the EDI;
* comorbidities are allowed except for those interfering with safety.

Exclusion Criteria:

* unable to respond to questions (parents or adolescents);
* no access to an Internet connection;
* insufficient mastery of Dutch language in parents or adolescents;
* physically incapable to work with the horses;
* unstable medication use;
* total intelligence quotient (IQ) equal to or below 80 on the Wechsler Intelligence Scale for Children (WISC-III-R or WISC-V);
* allergic or phobic to horses;
* insufficient regulation to safely handle the horses;
* therapy with horses within the last two years.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on the Emotion dysregulation Index (EDI) after start of the intervention | 3 times a week during 23 weeks from baseline
  The EDI-short form is a validated, change-sensitive, 13-item caregiver report measure of emotion regulation impairment for individuals who are at least 6 years of age. The scale used is Not at all=0, Mild=1, Moderate=2, Severe=3, or Very Severe=4. The EDI short form includes two scales: a 7-item Reactivity Index and a 6-item Dysphoria Index. Index raw scores will be converted into t-scores.

SECONDARY OUTCOMES:
Change from baseline of Quality of life as scored on the KIDSCREEN after 15 weeks and 1 year | The KIDSCREEN-27 will be assessed at baseline (T0), at week 2-6 (T1), at week17-23 (T2), week 25 (T3) and after 1 year (T4)
  The KIDSCREEN-27 is a generic health-related quality of life (HRQOL) questionnaire for children aged 8-18 years. There is a self-complete version (child and a proxy version (parent). It consists of 27 items measuring five dimensions: physical well-being, psychological well-being, parent relations & autonomy, social support & peers and school environment. Items are answered on a five-point Likert-type scale assessing frequency (never (1), seldom (2), sometimes (3), often (4), and always (5)) or intensity (not at all (1), slightly (2), moderately (3), very (4), and extremely (5)) with a one-week recall period. Negatively formulated items are recoded and the sum scores for respective dimensions are converted into T scores with a mean of 50 and a standard deviation (SD) of 10. Higher scores indicate better HRQOL.
Change from baseline of severity of autism spectrum symptoms as measured on the Social Responsiveness Scale (SRS-2) after 15 weeks and 1 year | The SRS-2 (parents) will be assessed at baseline (T0), at week 2-6 (T1), at week17-23 (T2), week 25 (T3) and after 1 year (T4).
  The Social Responsiveness Scale (SRS-2) measures deficits in social behavior associated with ASD and can be used to assess the severity of symptoms in ASD. The questionnaire will be completed by multiple raters (parents and teachers). The SRS-2 consists of 65 items scored in a Likert-like scale format ranging from not true=1, sometimes true=2, often true=3 to almost always true =4. It is designed to identify social impairment intrinsic to ASD and to quantify its severity across the duration of the treatment. A total score and five treatment subscale scores (Social Awareness; Social Cognition; Social Communication; Social Motivation; and Restricted Interests and Repetitive Behavior) are obtained. The accepted diagnostic criteria (cut point) for the SRS-2 for the association with a diagnosis of ASD are:<=59 (normal); 60-75 (mild to moderate ASD); and =>76 (severe ASD).
Change from baseline on the Goal Attainment Scale (GAS) after the intervention after 15 weeks | The GAS will be assessed in the fifth (week 7-11), tenth (week12-16) en fifteenth (week 17-23) sessions.
  Goal Attainment Scale is a method of scoring the extent to which the patient's individual goals are achieved in the course of the intervention. In effect, each patient has his own outcome measure, but this is scored in a standardized way as to allow statistical analysis. Each goal is rated on a six-point scale, capturing the degree of attainment for each goal area: The present situation is scored -2 (stable). When the patient improves, but achieves less than the expected level this is scored -1 and the expected level is scored 0. When he achieves a better than expected outcome this is scored +1 (somewhat better than the goal) or +2 (much better). Achieving a worse than expected outcome is scored -3 (somewhat worse) In this study, a maximum of 3-4 goals are identified, which are incorporated into a single GAS score.
Change from baseline of self-esteem as measured on the The Rosenberg Self-Esteem Scale (RSES) after 15 weeks and 1 year | Rosenberg Self-Esteem Scale will be assessed at the baseline (T0), at week 2-6 (T1), at week17-23 (T2), week 25 (T3) and after 1 year.
  The Rosenberg Self-Esteem Scale (RSES) [31] will be used to assess self-esteem. It is a widely used 10-item Likert-scale self-esteem measure. Items are answered on a four-point scale - ranging from strongly agree to strongly disagree - measuring positive and negative feelings towards the self. The Dutch version of the RSES is found to be a one-dimensional scale with high internal consistency and congruent validity and a Cronbach's alpha of 0.89
Change from baseline of Global functioning as measured on the Child Behavior Checklist (CBCL) after 15 weeks and 1 year | The whole version will be assessed at baseline, short version at week 2-6 (T1), at week17-23 (T2), week 25 (T3) and after 1 year (T4).
  For assessing emotional and/or behavioral problems we will use the CBCL/6-18, completed by parents , the TRF/6-18, completed by teachers, and the YSR/11-18, completed by youths. They include more than 100 items assessing behavioral and emotional problems that are answered on a three-point Likert-type scale (0 = not true, 1 = somewhat or sometimes true, 2 = very true or often true) by parents. The scores will display eight problem scales. The sum of the problem scales 1, 2 and 3 form the 'internalizing behavior' scale, whereas 7 and 8 form 'externalizing behavior'. All subscales together count for the total problem scale. T-scores are computed from raw scores; higher scores on the syndrome scales indicate a greater severity of problems. A T-score of 63 (90th percentile) demarcates the clinical range, which is an indication that a child needs professional help. For the competence scales, lower scores indicate greater severity. A T-score < 37 indicates the clinical range.
Change from baseline of Goal attainment as measured on the Outcome Rating Scale (ORS) after 15 weeks | The therapist will assess the SRS/ORS each session (week 3-23).
  For collecting client feedback we will use a brief questionnaires, the Outcome Rating Scale (ORS), which will be easily administered on a regular basis during treatment (https://www.scottdmiller.com/ scholarly-publications-handouts-vitae/).This allows treatment sessions to be evaluated at any time to ascertain whether or not individual treatments are 'on the right track' towards a successful outcome. The ORS is primarily focused on the well-being of the client and is administered at the beginning of the treatment session. The SRS is administered at the end of the session and deals with how the client has experienced the treatment session. The outcomes of the questionnaires are reflected in a graph on an iPad (or on paper when an iPad is not available) per interview to allow the height of the score and progress to be visualized during the sessions.
Change from baseline of family functioning as measured on the VGFO on T3 | This questionnaire will be assessed at the baseline (T0) and at week 25 (T3).
  Family functioning is assessed using a validated questionnaire: the Family Functioning Questionnaire (VGFO, 34 items) (https://www.praktikon.nl/wat-we-doen/vragenlijsten/vgo). The Family Functioning Questionnaire can be answered on a four-point scale ranging from 1 (not applicable) to 4 (completely applicable) with lower scores indicating more problems in family functioning.
Change from baseline of Global functioning as measured on the Teachers Report Form (TRF) after 15 weeks and 1 year | The whole version will be assessed at baseline, short version at week 2-6 (T1), at week17-23 (T2), week 25 (T3) and after 1 year (T4).
  For assessing emotional and/or behavioral problems we will use the TRF/6-18, completed by teachers. They include more than 100 items assessing behavioral and emotional problems that are answered on a three-point Likert-type scale (0 = not true, 1 = somewhat or sometimes true, 2 = very true or often true) by parents. The scores will display eight problem scales. The sum of the problem scales 1, 2 and 3 form the 'internalizing behavior' scale, whereas 7 and 8 form 'externalizing behavior'. All subscales together count for the total problem scale. T-scores are computed from raw scores; higher scores on the syndrome scales indicate a greater severity of problems. A T-score of 63 (90th percentile) demarcates the clinical range, which is an indication that a child needs professional help. For the competence scales, lower scores indicate greater severity. A T-score < 37 indicates the clinical range.
Change from baseline of Global functioning as measured on the Youth Self Report (YSR) after 15 weeks and 1 year | The whole version will be assessed at baseline, short version at week 2-6 (T1), at week17-23 (T2), week 25 (T3) and after 1 year (T4).
  For assessing emotional and/or behavioral problems we will use the YSR/11-18, completed by youths. They include more than 100 items assessing behavioral and emotional problems that are answered on a three-point Likert-type scale (0 = not true, 1 = somewhat or sometimes true, 2 = very true or often true) by parents. The scores will display eight problem scales. The sum of the problem scales 1, 2 and 3 form the 'internalizing behavior' scale, whereas 7 and 8 form 'externalizing behavior'. All subscales together count for the total problem scale. T-scores are computed from raw scores; higher scores on the syndrome scales indicate a greater severity of problems. A T-score of 63 (90th percentile) demarcates the clinical range, which is an indication that a child needs professional help. For the competence scales, lower scores indicate greater severity. A T-score < 37 indicates the clinical range.
Change from baseline of adherence as measured on the SRS after 15 weeks | The therapist will assess the SRS each session (week 3-23).
  For collecting client feedback we will use a brief questionnaires, the Session Rating Scale (SRS), which will be easily administered on a regular basis during treatment (https://www.scottdmiller.com/ scholarly-publications-handouts-vitae/).This allows treatment sessions to be evaluated at any time to ascertain whether or not individual treatments are 'on the right track' towards a successful outcome. The ORS is primarily focused on the well-being of the client and is administered at the beginning of the treatment session. The SRS is administered at the end of the session and deals with how the client has experienced the treatment session. The outcomes of the questionnaires are reflected in a graph on an iPad (or on paper when an iPad is not available) per interview to allow the height of the score and progress to be visualized during the sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Nanda Lambregt-Rommelse, Prof. Dr., Principal Investigator — Radboud/Karakter
Locations (3):
- Netherlands (3):
  - Karakter, Ede, Gelderland
  - Horses & Co, Heerjansdam
  - De Gagelhoeve, Mill

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trzmiel T, Purandare B, Michalak M, Zasadzka E, Pawlaczyk M. Equine assisted activities and therapies in children with autism spectrum disorder: A systematic review and a meta-analysis. Complement Ther Med. 2019 Feb;42:104-113. doi: 10.1016/j.ctim.2018.11.004. Epub 2018 Nov 5. PMID 30670226
- [Derived] den Boer JC, Klip H, Blonk A, Lenselink M, Kaijdoe SPT, Tielkes M, van Zandbeek A, Bres G, Herinx M, Staal WG, Rommelse N. Study Protocol: Pegasus: psychotherapy incorporating horses for 'therapy-resistant' adolescents with autism spectrum disorders, a study with series of randomised, baseline controlled n-of-1 trials. BMC Psychiatry. 2024 Jul 10;24(1):499. doi: 10.1186/s12888-024-05879-w. PMID 38987737

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT05200351/Prot_SAP_000.pdf